CLINICAL TRIAL: NCT01079975
Title: Predicting Factors for Depression in Patients With MS in Argentina
Brief Title: To Identify and Evaluate the Predictive Factors for Depression in Patients Diagnosed With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200077- 500
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Depression
MeSH Terms: conditions — Multiple Sclerosis; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, non controlled, multicentric, prospective study planned to be conducted in 350 subjects diagnosed with multiple sclerosis (MS) in 20 centres of Argentina to identify the predictive factors leading to depression. The incidence of depression symptoms and its influence in the evolution of the disease are unknown in the Argentinean population. Early diagnosis of depression symptoms allows the specific treatment of them and can also delay the rich apparition of the disease. This study intends to quantify the incidence of these symptoms and also aims to evaluate which are the predictive factors of the apparition of the depression.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic, demyelinating disease of the central nervous system and is considered to be one of the most common cause of neurological disability in young adults. The clinical and pathophysiological characteristics of the disease lead to the association of several conditions over time, among which the depression and/or the depression symptoms are one of the most important ones. The underlying mechanism of depression is not clear and the etiology of depression is considered to be multifactorial and especially associated to the psychosocial stress, to the presence of focal demyelinating lesions and to the immune malfunction. Several scales like Beck Depression Inventory Fast Screen (BDI FS), Mini Mental State Examination (MMSE), Hamilton Depression Rating Scale (HDRS) have been used to objectify the presence of depression symptoms in subjects with MS.

OBJECTIVES

Primary objective:

* Identification of the predictive factors for the development of depression symptoms in subjects with MS in Argentina

Secondary objective:

* Evaluation of the proportion of subjects that develop depression symptoms during the follow up

The subjects will be managed with the clinical and therapeutic elements that the treating doctors considered appropriate, without modifying their decisions due to the subjects' inclusion into the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 65 years of both sexes
* Subjects with established MS diagnosis according to the revised Mc Donald criteria - 2005 in any of its clinical forms
* Subjects with signed informed consent
* Subjects wiling to follow the study procedure

Exclusion Criteria:

* Subjects with diagnosis of depression at the moment of the initial evaluation
* Subjects receiving antidepressant drugs at the moment of the initial evaluation
* Subjects with moderate or severe cognitive impairment
* Antecedents of any other psychiatric disease
* Subjects that were receiving or have received any experimental treatment during the 6 months before the inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with diagnosed MS in Argentinean population.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Apparition and/or modification of depression symptoms through the agreed assessments | Each visit starting from the initial visit (Day 0) to end of the observation period (i.e. 24 months)
  The assessments will include Expanded Disability Status Scale, Hamilton Depression Rating Scale, Mini Mental State Examination, Beck Depression Inventory, clock drawing test and findings in magnetic resonance imaging.

SECONDARY OUTCOMES:
Proportion of subjects that developed depression symptoms during the study compared to the total population of subjects enrolled in the study | Initial visit (Day 0) to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Rey, Neurologist, Principal Investigator — Instituto de Investigacion Neurológica (Uruguay 840), Capital Federal City, Buenos Aires , 1015 , Argentina
Locations (1):
- Instituto de Investigacion Neurológica (Uruguay 840), Capital Federal, Buenos Aires, Argentina